CLINICAL TRIAL: NCT06933966
Title: ATTENUATION - A Multicenter Randomized Phase II Study of the Efficacy and Safety De-escalation Versus Standard Adjuvant Chemotherapy in Patients With Low Risk Localized Gastroesophageal Adenocarcinoma (PRODIGE99/FRENCH 39 Study)
Brief Title: Evaluation of Efficacy and Safety De-escalation Versus Standard Adjuvant Chemotherapy in Patients With Low Risk Localized Gastroesophageal Adenocarcinoma
Acronym: ATTENUATION
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Leon Berard (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ET23-350; 2023-509227-41-00 (EU CTIS Number)
Record Dates: First submitted 2025-03-21; First posted 2025-04-18 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Gastric Adenocarcinoma or Gastroesophageal Junction Adenocarcinoma or Esophageal Carcinoma; Non Metastatic Disease
Keywords: De-escalation post-operative chemotherapy; Gastric Adenocarcinoma or Gastroesophageal Junction Adenocarcinoma or Esophageal Adenocarcinoma
MeSH Terms: conditions — Esophageal Neoplasms; Adenocarcinoma Of Esophagus | interventions — Observation

STUDY DESIGN:
Intervention Model Description: Patients will be randomized according to the foloowing stratification criteria:
  * Primary tumour location (gastric vs gastro-esophageal junction and lower esophagus)
  * TRG score (Becker (B) or Mandard (M) classification): low (TRG 1a-b (B)/1-2 (M)) vs high (TRG 2-3 (B)/3-5 (M))
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental strategy: surveillance without FLOT post-operative chemotherapy (Experimental)
  Interventions: Other: observation alone
- Standard strategy : post-operative chemotherapy (4 cycles of FLOT) (No Intervention): Patients will received 4 cycles of FLOT after surgery.

INTERVENTIONS:
Other: observation alone — Patient will not received post-operative chemotherapy. There will be only surveillance until progression.
  Arms: Experimental strategy: surveillance without FLOT post-operative chemotherapy

SUMMARY:
The ATTENUATION study targets patients with gastric adenocarcinoma (GA), esophageal adenocarcinoma (EAC) or gastro-esophageal junction (GEJ) who have received 4 cycles of FLOT chemotherapy before the surgery. Standard post-operative management consists of chemotherapy with 4 cycles of FLOT.

However, the nature and duration of postoperative treatment are standardized and are not adapted to the specific tumor response of each patient. All patients are therefore referred to the same treatment regimen.

As a result, good responders (defined in particular by wide resection of the tumor and a good response to preoperative chemotherapy on the tumor removed during surgery) may be over-treated and exposed to unnecessary adverse events.

Only 50-60% of patients can start chemotherapy post-operatively, due to the potential residual adverse effects associated with surgery in particular. Thus, it would appear that preoperative chemotherapy is the most important factor in the overall efficacy of the treatment sequence. Moreover, numerous retrospective studies have reported a favorable outcome in patients with a major response to pre-operative treatment but who were unable to receive post-operative chemotherapy.

The hypothesis of this study is that surveillance after surgery in patients with gastric or gastroesophageal junction tumors, with a good response to preoperative chemotherapy could provide significant clinical benefit and favorable disease progression.

Participants will:

* be distributed in one of the two arms
* will be followed up every 3 months for 2 years, then every 6 months (clinical examination, imaging, quality-of-life questionnaire) subsequent years until 3 years after the randomization of the last patient.
* followed up until their death or their progression whether local, regional or metastatic.

ELIGIBILITY:
Inclusion Criteria:

* I1. Age ≥ 18 years, I2. Histologically proven non-metastatic (M0) gastric, oesophageal or gastroesophageal junction adenocarcinoma, I3. Subjects must have completed both pre-operative chemotherapy with a fluoropyrimidine-platinum containing regimen (FLOT 4 cycles) and microscopically complete (R0) resection prior to randomization.

Note for surgery: total or distal gastrectomy with D2 lymphadenectomy according to ESMO guidelines should have been completed for gastric and junctional Siewert type III cancers. Ivor Lewis oesophagectomy with two field lymphadenectomy should have been performed for junctional Siewert type I cancers and lower oesophageal adenocarcinomas. For Siewert type II cancers either total gastrectomy with D2-lymphadenectomy or oesophagectomy with two field lymphadenectomy should have been completed. Open, minimal invasive or hybrid surgical approaches are acceptable as long as the requirements above are fulfilled. In frail patients with Siewert I or II, transhiatal oesophagectomy with lymphadenectomy in the lower mediastinum without transthoracic access is acceptable. Regardless of the type of surgery a minimum of 16 (gastric cancer) or 7 lymph nodes (in case of oesophageal carcinoma) should have been resected and examined (ref TNM 8 eme edition)

I4. Low risk of disease recurrence, defined by the following criteria:

* Absence of lymph node involvement (ypN0), assessed on a min. of 16 or 7 lymph nodes according to the localization and,
* Either ypT0-2 (all TRG grade) or ypT3 (with TRG 1a-b according to Becker classification or TRG1-2 according to Mandard's classification), I5. ECOG Performance Status 0-1, I6. Patients fit to receive post-operative chemotherapy, I7. Interval between the date of surgery and the date of randomization no longer than 10 weeks, I8. Adequate organs function defined as : Absolute neutrophil count (ANC) ≥ 1.5 x 109/L; Platelets ≥ 100 x 109/L; Haemoglobin ≥ 9 g/dL (without transfusion within 7 days); Serum creatinine AND Calculated creatinine clearance as per MDRD or CKD-EPI formula ≤ 1.5 upper limit of normal (ULN) AND ≥ 40 mL/min /1.73m²; Serum total bilirubin ≤ 1.5 ULN OR Direct bilirubin ≤ ULN for patients with total bilirubin levels > 1.5 ULN (except for patients with Gilbert disease for whom a total serum bilirubin ≤ 3ULN is acceptable); AST and ALT ≤ 3 ULN; International Normalized Ratio (INR) and activated Partial Thromboplastin Time (aPTT)≤ 1.5 ULN .

I9. No contraindication to study assessments, I10. Signed and dated informed consent for prior to any study-specific procedure, I11. Women of childbearing potential accepting to use highly effective contraceptive measures or abstain from heterosexual activity, for the course of the study and at least an- 9 months after the end of the treatment with oxaliplatin - 6 months after the end of the treatment with fluorouracil - 2 months after the end of the treatment with docetaxel and men must use contraception during treatment and at least - 6 months after the end of the treatment with oxaliplatin, - 3 months after the end of the treatment with fluorouracil - 4 months after the end of the treatment with docetaxel.

I12. Patient must be covered by a medical insurance or equivalent.

Exclusion Criteria:

* E1. Oesophageal squamous cell carcinomas, E2. Tumour with Deficient MisMatch Repair (MMR) and/or Microsatellite Instability status, E3. Dihydro Pyrimidine Dehydrogenase (DPD) deficiency, NB: if not previously done, the following blood chemistry level must be perform at screening, : blood uracil level - uracilemia dosing result is mandatory prior the inclusion E4. Persistent toxicities related to prior treatment of grade>1, E5. QTcF longer than 450 msec for men and longer than 470 msec for women, E6. Hypokalemia OR Hypomagnesemia OR Hypocalcemia Grade>1

E7. Contraindication to postoperative treatment (FLOT):

* Known history of hypersensitivity to fluorouracil, oxaliplatin, docetaxel or calcium folinate to any of their excipients, according to the SmPCs of these products OR
* Peripheral sensory neuropathy with functional impairment prior to first treatment according the SmPC of oxaliplatin OR
* Clinically significant active heart disease or myocardial infarction within 6 months OR
* Recent or concomitant treatment with brivudine or recent treatment with live vaccines (minimal wash out period before randomisation: 4 weeks) E8. Any concurrent chemotherapy, Investigational product for cancer treatment. E9. Concurrent enrolment in another clinical study, unless it is an observational (non-interventional) clinical study E10. Suspicion of serious infection, E11. Pregnant or breastfeeding woman, E12. Patient under tutorship or curatorship of deprived of liberty.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2030-09-01 (Estimated); Study Completion 2032-09-01 (Estimated)

PRIMARY OUTCOMES:
3 year Overall Survival rate | From the date of randomisation to 3 years post-randomisation follow-up visit.
  The primary endpoint will the 3-year Overall Survival (OS) rate, described as the proportion of patients still alive 3 years after the date of randomization.
3 year disease-free survival rate | Time from the date of randomisation to 3 year post-randomisation follow-up visit
  The co-primary endpoint is the 3-year Disease-Free Survival rate, considered as a binary variable with a success defined as being relapse-free at 3 years.

SECONDARY OUTCOMES:
Overall survival | Time from the date of randomisation to the date of death due to any cause or to the date of last contact if patient is still alive (censored patients), assessed up to 60 months.
  The overall survival (OS) will be defined as the time from the date of randomization to the date of death due to any cause or to the date of last contact if patient is still alive (censored patients).
Disease-Free Survival (DFS) | From the date of randomization to the date of the first documented relapse of the disease or death due to any cause, whichever occurs first, assessed up to 60 months.
  The Disease-Free Survival (DFS) will be defined as the time from the date of randomization to the date of the first documented relapse of the disease or death due to any cause, whichever occurs first. Patients alive and disease-free at the time of the analysis will be censored at the date of their last tumoral evaluation.
Type of Relapses | From the date of randomization to the date of the first documented relapse of the disease, assessed up to 60 months.
  The relapses will be described by their location (either locoregional or distant relapse).
The tolerability profile | From date of randomization to 3 years follow-up visit or death due to any cause, whichever came first, assessed up to 60 months
  The tolerability profile will be assessed continuously using the NCI-CTC AE version 5.0. All Adverse Events (AE), whichever their relationship with study treatments, all Serious AE, all Suspected Unexpected Serious Adverse Reactions and all toxic deaths, will be reported.
The health-related quality of life by QLQ-C30 | At Baseline and every year after randomisation during 3 years.
  The health-related quality of life will be assessed using the EORTC Quality of Life Questionnaire (QLQ-C30). Descriptive statistics and graphs will be reported to evaluate Quality of life in the 2 study arms. Mixed model for repeated measure and time to deterioration will be used to analyse longitudinal Quality of life.
The nutritional status by food intake changes | At baseline, every 3 months visits during the first 2 years then every 6 months until 3 years post-randomisation.
  The nutritional status will be assessed at baseline and during the course of treatment by a descriptive analysis of food intake changes.
ctDNA positivity | At baseline, every 3 months visits during the first 2 years then every 6 months until 3 years post-randomisation.
  The ctDNA positivity will be described in each arm in terms of proportion of positivity at each time point and delay between ctDNA positivity and recurrence documented on imaging.
The feasibility of using a standardized pathological report | At baseline visit only
  The feasibility of using a standardized pathological report will be described in the whole study population by the adherence to the standardized report (proportion of patients with a report and quality of filling).
The health-related quality of life by QLQ-OG25 | At Baseline and every year after randomisation during 3 years.
  The health-related quality of life will be assessed using the Gastric Cancer module (EORTC QLQ-OG25). Descriptive statistics and graphs will be reported to evaluate Quality of life in the 2 study arms. Mixed model for repeated measure and time to deterioration will be used to analyse longitudinal Quality of life.
The nutritional status by sarcopenia | At baseline, every 3 months visits during the first 2 years then every 6 months until 3 years post-randomisation.
  The nutritional status will be assessed at baseline and during the course of treatment by a descriptive analysis of sarcopenia. It will be analysed with muscle mass evaluation (computed tomography scans at lumbar level 3).
The physical performance | At baseline, every 3 months visits during the first 2 years then every 6 months until 3 years post-randomisation.
  The physical performance will be assessed at baseline and during the course of treatment by a descriptive analysis of handgrip test.
The nutritional status by systemic inflammation (CRP) | At baseline, every 3 months visits during the first 2 years then every 6 months until 3 years post-randomisation.
  The nutritional status will be assessed at baseline and during the course of treatment by a descriptive analysis of measurements of serum C-reactive protein (CRP).
The nutritional status by measurements of albumin | At baseline, every 3 months visits during the first 2 years then every 6 months until 3 years post-randomisation.
  The nutritional status will be assessed at baseline and during the course of treatment by a descriptive analysis of measurements of albumin.
The nutritional status by weight changes | At baseline, every 3 months visits during the first 2 years then every 6 months until 3 years post-randomisation.
  The nutritional status will be assessed at baseline and during the course of treatment by a descriptive analysis of weight changes.
The nutritional status by body mass index evaluation | At baseline, every 3 months visits during the first 2 years then every 6 months until 3 years post-randomisation.
  The nutritional status will be assessed at baseline and during the course of treatment by a descriptive analysis of body mass index (BMI) evaluation.

CONTACTS AND LOCATIONS:
Overall Officials: Christelle DE LA FOUCHARDIERE, MD, Principal Investigator — Institut Paoli-Calmettes, Department of Medical Oncology
Locations (3):
- France (3):
  - Centre Léon Bérard, Lyon
  - Institut Paoli-Calmettes, Marseille
  - AP-HP - Hôpital Saint-Antoine, Paris